CLINICAL TRIAL: NCT02169271
Title: A Randomized Phase II Trial of Low Dose Aspirin Versus Placebo in High-Risk Individuals With CT-Detected Subsolid Lung Nodules
Brief Title: Acetylsalicylic Acid Compared to Placebo in Treating High-Risk Patients With Subsolid Lung Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-01311; NCI-2014-01311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IEO-833/13F; HHSN261201200034I; EIO 833/13F; 2013-004862-32; TO-RFP A; N01-CN-2012-00034; IEO 833/13F (IEO37); MDACC: 2013-0732; IEO 37; 2013-0732 (Other: M D Anderson Cancer Center); MDA2013-01-01 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH); NCT02135497 (obsolete NCT alias)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Current Smoker; Former Smoker; Multiple Pulmonary Nodules; Tobacco Use Disorder
MeSH Terms: conditions — Smoking Cessation; Multiple Pulmonary Nodules; Tobacco Use Disorder | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (acetylsalicylic acid) (Experimental): Patients receive acetylsalicylic acid PO QD for 12 months.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 12 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm I (acetylsalicylic acid)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies acetylsalicylic acid compared to placebo in treating high-risk patients with subsolid lung nodules. A nodule is a growth or lump that may be malignant (cancer) or benign (not cancer). Chemoprevention is the use of drugs to keep cancer from forming or coming back. The use of acetylsalicylic acid may keep cancer from forming in patients with subsolid lung nodules.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The evaluation of the effect of aspirin (acetylsalicylic acid) as a chemopreventive agent for lung cancer.

SECONDARY OBJECTIVES:

I. The modulation of biological markers after treatment and the correlation of these findings with modification of lung nodules diameters.

II. The per-lesion analysis including the evaluation of lung nodule density before and after treatment, the number and size of non target lesions including solid nodules and evaluation of response according to modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive acetylsalicylic acid orally (PO) once daily (QD) for 12 months.

ARM II: Patients receive placebo PO QD for 12 months.

After completion of study treatment, patients are followed up for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic current or former smokers (having stopped within the last 20 years)
* Smoking history >= 20 pack/years; subjects must be included in an ongoing annual screening with low dose CT scan or must have two consecutive CT outside the context of a screening program confirming subsolid nodules
* Subjects must have subsolid (non solid or partially solid) nodules with size between 4 and 10 mm with any volume doubling time (VDT) not candidate to surgical excision and/or subsolid (non solid or partially solid) nodule larger than 10 mm with VDT higher than 400 days and not candidate to surgical excision
* All nodules should be persistent at least after three months follow up with 1 dimension (1d)-CT; a reduction up to 15% of the diameter of the largest target nodule from the previous CT scan is allowed
* All current smokers should accept to receive support for smoking cessation
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) and/or history of Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional ULN
* Serum creatinine =< institutional ULN
* Women of child-bearing potential (from first menstruation to 1 year after last menstruation) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Signed informed consent

Exclusion Criteria:

* Subjects with chronic treatment (at least twice/week for more than 3 months) with aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
* History of allergic reactions attributed to compounds of similar chemical or biological composition to aspirin, NSAIDs, cyclooxygenase-2 (COX2) inhibitors
* Invasive malignancy (with the exclusion of basal cell carcinoma or skin squamous cell carcinoma) diagnosed during the last 2 years before randomization; stage I-II invasive malignancies that were diagnosed more than 2 years prior to randomization and have been treated curatively are allowed as long as all treatment is finished at least 18 months prior to randomization
* History of therapeutic doses of anticoagulants including warfarin and low molecular weight heparin (e.g. for prior deep venous thrombosis and pulmonary embolisms) in the preceding year
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with aspirin
* Individual may not be receiving any other investigational agents, antiplatelet agents (e.g. aspirin, clopidogrel [Plavix or others]), anticoagulants (e.g. heparin or heparinoids, Coumadin, or others), methotrexate, lithium
* Participants with bleeding diathesis, history of gastric/duodenal ulcers in the last 5 years, NSAID-precipitated bronchospasm, patients unwilling or unable to limit alcohol consumption to i.e. =< 3 alcohol drinks a day
* Participants who in the opinion of the principal investigator (PI) will be at higher risk of acetylsalicylic acid (ASA)-related complications
* Participants with known inability to adequately absorb oral medication

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Bonanni, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- M D Anderson Cancer Center, Houston, Texas, United States
- European Institute of Oncology, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 619 ld-CT scans, belonging to the lung screening programs, showed potentially eligible nodules. A total of 109 subjects signed a written informed consent and underwent baseline visit while 98 have been randomized.
Pre-assignment Details: After enrollment, 11 participants were not randomized (baseline screening failures)
Groups:
- Aspirin: 1 tablet of aspirin 100 mg a day for one year
- Placebo: 1 tablet of placebo a day for one year
Period: Overall Study
Arm/Group | Aspirin | Placebo
Started | 49 | 49
Completed | 48 | 47
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (4.1) | 64.6 (4.7) | 64.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 21 | 22 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 0 | 1
  Italy | 48 | 49 | 97
Sum of longest diameters of baseline target nodules [Mean (Standard Deviation); unit: millimeters] | 8.5 (4.3) | 11 (11.3) | 9.8 (8.6)
Sum of diameters of baseline target nodules [Mean (Standard Deviation); unit: millimeters] | 6.8 (2.8) | 7.2 (2.7) | 7.0 (2.8)
Baseline lesion volume [Mean (Standard Deviation); unit: Millimeter^3] | 138 (139) | 151 (151) | 145 (145)
Baseline lesion density [Mean (Standard Deviation); unit: Hounsfield Unit] | -628 (76) | -663 (98) | -647 (90)
Circulating biomarkers and miRNA risk score [Mean (Standard Deviation); unit: Score on a scale] — Scale from -20 to +30 which measure the risk of lung cancer. Higher values indicate higher risk. A value<0 is considered negative, a value ≥0 positive for lung cancer.
  Score on a scale | 10.4 (9.5) | 10 (10.6) | 10.2 (10)
Circulating Thromboxane [Mean (Standard Deviation); unit: ng/mL] | 60.4 (32.6) | 61.1 (37.3) | 60.8 (34.8)
Circulating Prostaglandin E metabolite (PGEM) normalized to uCr concentration [Mean (Standard Deviation); unit: pg/mg creatinine] | 385 (218) | 334 (213) | 359 (216)
Circulating Leukotriene E4 normalized to uCr concentration [Mean (Standard Deviation); unit: pg/mg creatinine] | 1701 (1670) | 1226 (909) | 1463 (1359)
Circulating High sensitive CRP [Mean (Standard Deviation); unit: mg/dL] | 0.47 (1.01) | 0.29 (0.52) | 0.38 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Sum of Longest Diameters of Baseline Target Nodules (Person-specific Analysis)
Description: Difference (12 month-baseline) in the sum of longest diameters of baseline target nodules.
Time Frame: Twelve-month treatment
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
millimeter (mm) | 0.3 (2.54) | -0.12 (1.55)

2. Secondary Outcome: Change in the Sum of Baseline Target Nodules Diameters (Per Nodules Analysis)
Description: Difference (12 month-baseline) in the sum of baseline target nodules diameters
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
millimeter (mm) | 0.1 (2.4) | -0.1 (1.1)

3. Secondary Outcome: Change in Lesion Volume
Description: Difference (12 month-baseline) in lesion volume
Time Frame: Baseline to 1 year
Measure: Mean (Standard Deviation); unit: millimiter^3 (mm3)
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
millimiter^3 (mm3) | -4.5 (78) | -4.8 (134)

4. Secondary Outcome: Change in Lesion Density
Description: Difference (12 month-baseline) in lesion density
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: Hounsfield unit (HU)
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
Hounsfield unit (HU) | 24 (65) | 28 (78)

5. Secondary Outcome: Modulation of Thromboxane B2
Description: Difference (12 month-baseline) in biomarker concentration
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
ng/mL | -35.8 (53.4) | 20.5 (50.7)

6. Secondary Outcome: Modulation of Prostaglandin E Metabolites (Normalized to Urinary Creatinine Concentration)
Description: Difference (12 month-baseline) in biomarker concentration
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
pg/mg creatinine | -60.7 (210) | 29.8 (215)

7. Secondary Outcome: Modulation of Leukotriene E4 (Normalized to Urinary Creatinine Concentration)
Description: Difference (12 month-baseline) in biomarker concentration
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
pg/mg creatinine | -235 (1240) | -9 (592)

8. Secondary Outcome: Modulation of High Sensitive CRP
Description: Difference (12 month-baseline) in biomarker concentration
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
mg/dL | -0.12 (0.88) | -0.08 (0.5)

9. Secondary Outcome: Modulation of miRNA Prediction Risk Score
Description: Difference (12 month-baseline) of the score on a scale (scale from -20 to +30 which measure the risk of lung cancer. Higher values indicate higher risk. A value<0 is considered negative, a value ≥0 positive for lung cancer).
Time Frame: Baseline up to 1 year
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Aspirin | Placebo
Number analyzed (Participants) | 49 | 49
Score on a scale | 0.14 (8.94) | 0.36 (7.36)

ADVERSE EVENTS:
Time Frame: Baseline up to 13 months
Arm/Group | Aspirin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 8/49 | 4/49
Other Adverse Events (participants affected / at risk) | 43/49 | 41/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=49) | Placebo (N=49)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Balanitis (Infections and infestations) | 1 (1) | 0 (0)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Increased volume of target lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Neoplasms benign, malignant and unspecified (including cuysts and polyps)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal fissures (Surgical and medical procedures) | 1 (1) | 0 (0)
Penile implant (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin (N=49) | Placebo (N=49)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Vitreous hemorrage (Eye disorders) | 0 (0) | 1 (1)
Other (Eye disorders) | 2 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Lower gastrointestinal hemorrage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 4 (5) | 3 (6)
Hemorroidal hemorrage (Gastrointestinal disorders) | 2 (2) | 2 (6)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 5 (5)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorroids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder, other (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flu-like symptoms (General disorders) | 5 (5) | 7 (8)
Localized edema (General disorders) | 1 (1) | 0 (0)
Non-cardia chest pain (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 3 (6) | 4 (4)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 10 (18) | 5 (10)
Urinary tract infection (Infections and infestations) | 4 (8) | 0 (0)
Tooth infection (Infections and infestations) | 2 (2) | 2 (2)
Penile Infection (Infections and infestations) | 1 (1) | 0 (0)
Laryingitis (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Other (Infections and infestations) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Bilirubin increased (Investigations) | 2 (2) | 2 (2)
Other (Investigations) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 7 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 7 (10) | 4 (12)
Paresthesia (Nervous system disorders) | 2 (5) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Other (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Other (Psychiatric disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 4 (6)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal hemorrage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vagynal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (9)
Epistaxix (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 7 (8)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sore theroat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Other (Surgical and medical procedures) | 4 (5) | 4 (4)
Hematoma (Vascular disorders) | 2 (3) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 3 (18)
Other (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT02169271/Prot_SAP_ICF_000.pdf